CLINICAL TRIAL: NCT06391489
Title: Piloting A Telehealth Deliverable Self-Management and Cognitive Training Program (HOBSCOTCH, HOme Based Self-Management and COgnitive Training CHanges Lives) for People With Post Acute COVID-19 Syndrome (PACS)
Brief Title: HOBSCOTCH for People With Post Acute COVID-19 Syndrome (PACS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Elaine T. Kiriakopoulos, Assistant Professor of Neurology, Geisel School of Medicine at Dartmouth Director, HOBSCOTCH Institute for Cognitive Health & Well-Being Dartmouth Hitchcock Epilepsy Center, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY 02002402
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Post Acute COVID 19 Syndrome; Memory Impairment; Memory Dysfunction; Cognitive Dysfunction
Keywords: Post Acute COVID 19 Syndrome; Long COVID; Memory; Cognitive Training; Self-Management
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Memory Disorders; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PACS Participant With Cognitive and Memory Dysfunction (Other): Participants will receive the HOBSCOTCH-PACS intervention consisting of 1:1 sessions delivered once per week including:
  1 pre-HOBSCOTCH Session (on webcam or by phone)
  1 educational session (on webcam) 6 HOBSCOTCH intervention sessions (webcam or phone)
  1 wrap-up session (webcam or phone)
  Interventions: Behavioral: HOBSCOTCH-PACS

INTERVENTIONS:
Behavioral: HOBSCOTCH-PACS — HOme-Based Self-management and COgnitive Training CHanges lives (HOBSCOTCH) HOBSCOTCH is a home-based self-management program to treat cognitive symptoms and improve quality of life, while minimizing the barriers of access to care. The program is based on Problem Solving Therapy (PST) and teaches problem solving strategies and compensatory mechanisms to help manage cognitive dysfunction and enhance quality of life. HOBSCOTCH-PD is an adaptation of the HOBSCOTCH program for people with PD and incorporates education about Parkinson Disease and cognition into the education module.

SUMMARY:
The goal of this pilot study is to assess the feasibility of adapting and delivering the existing home-based epilepsy self-management intervention, HOBSCOTCH, for people with Post Acute Covid Syndrome (PACS).

The main questions it aims to answer are:

Can the current HOBSCOTCH program be adapted for people with PACS?

Will people with PACS experience improved quality of life similar to that found in people with epilepsy after participating in the HOBSCOTCH program?

Participants will be asked to:

* attend nine, one-hour virtual (online and/or by telephone) HOBSCOTCH-PACS sessions with a one-on-one certified HOBSCOTCH-PACS coach
* complete a brief clinical questionnaire about their diagnosis of PACS
* complete seven questionnaires before and after the HOBSCOTCH-PACS sessions about their quality of life, memory and thinking processes (objective and subjective cognition), about their physical and mental health and about autonomic symptoms associated with their diagnosis of PACS
* keep a short daily diary (using a smart phone app or on paper) about their PACS symptoms and use of the self-management strategies taught in the HOBSCOTCH-PACS program
* complete two brief surveys to assess satisfaction with their experience after the entire HOBSCOTCH-PACS program

ELIGIBILITY:
Inclusion Criteria:

* Literate, English-speaking with grade 12 or equivalent in education
* Self-reported diagnosis of PACS
* Self-reported cognitive/memory difficulties
* Telephone and internet access

Exclusion Criteria:

* Cognitive dysfunction that precludes participation in giving informed consent
* Significant visual impairment precluding reading or writing
* No reliable telephone or internet access
* Neurodegenerative illness (i.e. dementia)
* Acute psychiatric disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in overall quality of life as measured by comparing PROMIS-10 Global Health scores pre- and post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  PROMIS Global-10 is a validated 10-question survey and part of the Patient-Reported Outcomes Measurement Information System (PROMIS) used to assess health care-related quality of life. Measures include overall health, pain, fatigue, social health, mental health, and physical health. 9 of the items are scored on a Likert Scale of 1 - 5 with 5 representing the best health care-related quality of life; higher scores are associated with better quality of life. One item related to pain is measured on a scale of 1 - 10 with 10 being the worst possible pain.
Change in subjective cognition as measured by comparing Neuro-QOL Item Bank v2.0 Cognitive Function scores pre- and post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  The Cognitive Function sub-scale of the Neuro-QOL is a brief validated tool developed by the NIH for use in patients with neurological disease. Scores range from 8 to 40, with a higher score indicating better reported cognitive functioning.

SECONDARY OUTCOMES:
Change in objective cognition as measured by comparing Symbol-Digit Modalities Test scores pre- and post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  The Symbol Digit Modalities Test (SDMT) is a validated tool that measures cognitive processing speed. It requires a person to substitute a number (1 - 9), either orally or written, for randomized presentations of geometric figures over 90 seconds. Scores range between 0 and 100 with a lower score representing poorer performance.
Change in objective cognition as measured by comparing California Verbal Learning Test-III scores pre- and post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  The California Verbal Learning Test-III is a validated verbal learning and memory assessment. It consists of a 16-word, list-recall task with up to five learning/recall trials. Higher scores of recall over time are associated with better performance.
Change in objective cognition as measured by comparing Montreal Cognitive Assessment (MOCA) scores pre- and post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  The Montreal Cognitive Assessment (MOCA) is a validated 30 item test that helps healthcare professionals detect cognitive impairments. The test examines seven domains (aspects) of cognitive function with a total of 11 different exercises and tasks including: executive and visuospatial function, naming, attention, language, abstraction, delayed recall, orientation.
  Scores range from 0 - 30 with higher scores indicating less cognitive impairment.
Change in self-reported autonomic symptoms as measured by comparing COMPASS-31 scores pre- and post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  COMPASS 31 is an abbreviated quantitative measure of autonomic symptoms based on the 169-item Autonomic Symptom Profile (ASP) and its validated 84-question scoring instrument, the Composite Autonomic Symptom Score (COMPASS). The six domain scores sum to a total COMPASS 31 score of 0 to 100, and a higher COMPASS 31 score indicates more severe autonomic symptoms.
Change in subjective physical and mental health as measured by comparing PROMIS-29+2 scores pre- and post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  PROMIS-29+2 is part of the Patient-Reported Outcomes Measurement Information System (PROMIS). It assesses pain intensity and seven health domains: physical functioning, fatigue, pain interference, depression, anxiety, social participation, and sleep disturbance in addition to two (+2) subjective cognition questions. The test is scored on a 5-point Likert scale, except for one question on subjective pain that uses a scale of 1 - 10. The domains are scored separately and compared to a mean score. Scores below 1 SD above the mean do not represent a problem for the person, or perhaps a mild concern. Between 1 and 2 SD reflect a moderate concern or interference in day to day function. Scores worse than 2SD beyond the mean score are considered to reflect poorer subjective physical or mental health.
Change in participants' self-reports of mood as measured by comparing scores on the PHQ-8 pre- and post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  The PHQ-8 is a self-reported, standardized set of 8 questions used to assess the presence and severity of depression symptoms. It is a shortened version of the PHQ-9, omitting the last question about suicidal thoughts or self-harm. The items are scored on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). Higher scores are consistent with greater symptoms of poor mood or depression.
Change in participants' self-reports of anxiety as measured by comparing scores on the GAD-7 pre- and post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  The Generalized Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for measuring symptoms of generalized anxiety disorder (GAD). The seven items are scored on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). Higher scores suggest greater symptoms of anxiety.
Changes in brain fog symptoms as measured by comparing daily self-reported symptoms pre- and post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  Participants will self-report their brain fog symptoms using a smartphone app or paper log. The smart phone app was developed by the HOBSCOTH program at Dartmouth-Hitchcock and is used clinically in the HOBSCOTCH program.
Changes in autonomic symptom frequency as measured by comparing daily self-reported symptoms pre- and post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  Participants will self-report their autonomic symptom frequency using a smartphone app or paper log. The smart phone app was developed by the HOBSCOTH program at Dartmouth-Hitchcock and is used clinically in the HOBSCOTCH program.
Changes in participants' use of memory strategies as measured by a daily self-reported diary compared at baseline/pre-HOBSCOTCH-PACS and post-HOBSCOTCH-PACS intervention. | Recorded daily and compared between baseline/pre-HOBSCOTCH-PACS and post-HOBSCOTCH-PACS intervention.
  Participants will self-report their use of the memory strategies they learn in the HOBSCOTCH-PACS program using a smartphone app developed by the HOBSCOTH program at Dartmouth-Hitchcock or in a paper log.
Changes in participants' self-reports of wellbeing as measured by comparing daily reports of well-being at baseline/pre-HOBSCOTCH-PACS and post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  Participants will self-report daily well-being information on a single item Likert-scale of well-being throughout the entire study by use of a smartphone app developed by the HOBSCOTH program at Dartmouth-Hitchcock or in paper log.
Evaluation of participants' engagement and compliance in HOBSCOTCH-PACS by measuring completed HOBSCOTCH sessions and use of smart phone app/daily diary from baseline (pre-HOBSCOTCH-PACS) through post-HOBSCOTCH-PACS intervention. | Baseline (pre-HOBSCOTCH-PACS) and post-HOBSCOTCH-PACS, approximately 9 weeks later.
  Participants' completed HOBSCOTCH-PACS sessions and smart phone app/daily diary logs will be assessed and recorded weekly. Greater number of sessions and daily diary records indicate better engagement and compliance.
Evaluation of participant satisfaction with the HOBSCOTCH-PACS intervention as measured by Satisfaction for PTE Participants as measured by analyzing a Participant Satisfaction Survey at the end of the study. | After completion of the HOBSCOTCH-PACS intervention and all post-HOBSCOTCH-PACS assessments, approximately 9 weeks after enrollment.
  The Participant Satisfaction Survey has been developed through the original HOBSCOTH Institute at Dartmouth and is used in clinical practice for program evaluation and quality improvement. It contains 9 items scored on a 5-point Likert scale with a higher score indicating greater satisfaction with the program. Four open-ended questions exist for participants to express likes, dislikes, areas for improvement and additional comments.
Evaluation of participants' perception of shared-decision making during HOBSCOTCH-PACS intervention as measured by CollaboRATE score. | After completion of the HOBSCOTCH-PACS intervention and all post-HOBSCOTCH-PACS assessments, approximately 9 weeks after enrollment.
  CollaboRATE is a brief patient survey focused on shared decision making. It employs a 3-item assessment of patient perception of how much effort was made to hear, understand and incorporate their concerns into the program. The items are measured on a 10-point Likert scale in which 0 indicates that no effort was made and 9 indicates every effort was made. Higher scores indicate a greater degree or positive impression of patient perception of shared decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine T Kiriakopoulos, MD, MPH, MSc, Principal Investigator — Dartmouth-Hitchcock, Dartmouth College
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No